CLINICAL TRIAL: NCT01213251
Title: Post-Myocardial Infarction Remodeling Prevention Therapy
Acronym: PRomPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRomPT
Record Dates: First submitted 2010-09-28; First posted 2010-10-01 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction; Pacing Therapy; Cardiac Remodeling; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single Site Pacing (Experimental)
  Interventions: Device: Single Site Pacing
- Dual Site Pacing (Experimental)
  Interventions: Device: Dual Site Pacing
- Control (No Intervention)

INTERVENTIONS:
Device: Single Site Pacing — Subjects will be implanted with a CRT-D that delivers pacing via the Left Ventricular lead.
  Arms: Single Site Pacing
Device: Dual Site Pacing — Subjects will be implanted with a CRT-D that delivers pacing via the Left Ventricular and Right Ventricular lead.
  Arms: Dual Site Pacing

SUMMARY:
The purpose of this study is to demonstrate the feasibility of pacing as a therapy to prevent adverse remodeling of the myocardium following an acute myocardial infarction (MI) in patients at highest risk for adverse myocardial remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial Infarction (MI) within the past 10 days
* Peak Creatine Phosphokinase (CPK) greater than 3000 Units/Litre (U/L) at time of MI, or a troponin T (TnT) greater than 10 micrograms/Litre (mcg/L)
* At least 18 years old
* Willing to comply with the protocol

Exclusion Criteria:

* Documented MI greater than 10 days
* Chronic renal disease, as defined by estimated glomerular filtration rate (eGFR) less than 30 milliliters/minute/1.73 square meter
* Life expectancy less than 18 months, as determined by a physician
* Existing pacemaker, Implantable Cardioverter Defibrillator (ICD), or Cardiac Resynchronization Therapy (CRT) device
* QRS duration greater than 120 milliseconds (ms)
* Coronary Artery Bypass Graft (CABG) within 30 days prior to MI, or CABG procedure planned
* Third degree atrioventricular (AV) block or symptomatic bradyarrhythmia
* Persistent atrial fibrillation (AF) that is not self terminating within 7 days or is terminated electrically or pharmacologically
* Permanent AF that is non self terminating, with cardioversion failed or not attempted within the past year
* New York Heart Association (NYHA) Class IV
* Non-ischemic cardiomyopathy
* Pregnant or planning to become pregnant during the study
* Enrolled or planning to participate in a concurrent drug and/or device study during the course of this clinical trial. Co-enrollment in concurrent trials is only allowed with documented pre-approval from Medtronic, documenting that there is not a concern that co-enrollment could confound the results of this trial.
* Breast feeding
* Of a vulnerable population as determined by local law or requirement, or a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-12; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, MD, Principal Investigator — Columbia University; Angel Leon, MD, Principal Investigator — Emory University
Locations (26):
- United States (17):
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Kaiser Permanente, Los Angeles, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Lexington Cardiac Research Foundation, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Carolina Heart Specialists, Gastonia, North Carolina
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Chattanooga Heart Institute, Chattanooga, Tennessee
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Saint Thomas Research Institute, LLC, Nashville, Tennessee
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Delgado Cardiovascular Associates, Houston, Texas
  - Spokane Cardiology, Spokane, Washington
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hôpital Cardiologique du Haut-Lévêque, Bordeaux-Pessac
  - Centre Hospitalier Régional Universitaire de Lille, Lille
- Germany (2):
  - Herzzentrum Leipzig GmbH, Leipzig
  - University Hospital Mannheim, Mannheim
- Hungary (2):
  - Maygar Honvédség Honvédkorház, Budapest
  - Semmelweis University Heart Center, Budapest
- Prince Salman Heart Centre, King Fahad Medical City, Saudi Arabia
- Vychodoslovensky ustav srdcovych a cievnych chorob, a.s., Košice, Slovakia

REFERENCES:
- [Derived] Stone GW, Chung ES, Stancak B, Svendsen JH, Fischer TM, Kueffer F, Ryan T, Bax J, Leon A; PRomPT Trial Investigators. Peri-infarct zone pacing to prevent adverse left ventricular remodelling in patients with large myocardial infarction. Eur Heart J. 2016 Feb 1;37(5):484-93. doi: 10.1093/eurheartj/ehv436. Epub 2015 Aug 30. PMID 26321236
- See also: The Post-Myocardial Infarction Pacing Remodeling Prevention Therapy (PRomPT) Trial: Design and Rationale — http://dx.doi.org/10.1016/j.cardfail.2015.03.005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients exited study prior to randomization.
Groups:
- Single Site Pacing: Subjects randomized to the group that will be implanted with a CRT-D that delivers pacing via the Left Ventricular lead.
- Dual Site Pacing: Subjects randomized to the group that will be implanted with a CRT-D that delivers pacing via the Left Ventricular and Right Ventricular lead.
- Control: Subjects randomized to the group that will not have a device implanted and will be managed according to conventional medical management.
Period: Overall Study
Arm/Group | Single Site Pacing | Dual Site Pacing | Control
Started | 40 | 41 | 45
Completed | 34 (Patients that had the 18-Month follow-up visit) | 37 (Patients that had the 18-Month follow-up visit) | 34 (Patients that had the 18-Month follow-up visit)
Not Completed | 6 | 4 | 11
Not completed — Death | 2 | 1 | 2
Not completed — Exit | 3 | 2 | 8
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Missed 18-Month Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Site Pacing | Dual Site Pacing | Control | Total
Number analyzed (Participants) | 40 | 41 | 45 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10) | 60 (12) | 54 (11) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 12 | 33
  Male | 28 | 32 | 33 | 93
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 0 | 1
  Black or African American | 3 | 3 | 5 | 11
  Hispanic or Latino | 0 | 1 | 3 | 4
  White or Caucasian | 19 | 16 | 18 | 53
  Not reportable per local laws or regulations | 18 | 20 | 19 | 57
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28 (6) | 30 (5) | 29 (4) | 29 (5)
Systolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 114 (16) | 118 (21) | 119 (17) | 117 (18)
Diastolic Blood Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 73 (11) | 71 (12) | 74 (11) | 73 (11)
Heart Rate from Physical Exam (BPM) [Mean (Standard Deviation); unit: BPM] | 80 (15) | 80 (13) | 79 (14) | 79 (14)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 43 (9) | 43 (10) | 45 (9) | 44 (9)
Left Ventricular End Diastolic Volume (LVEDV) [Mean (Standard Deviation); unit: mL] | 107 (25) | 107 (31) | 116 (29) | 111 (29)
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: mL] | 62 (23) | 62 (22) | 65 (24) | 63 (23)
QRS Width (msec) [Mean (Standard Deviation); unit: msec] | 94 (17) | 97 (17) | 88 (13) | 93 (16)
NYHA [Number; unit: participants] — The New York Heart Association (NYHA) score classifies patients' heart failure according to the severity of their symptoms. In particular, Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Unable to carry on any physical activity without discomfort.
  participants
    I | 9 | 12 | 11 | 32
    II | 10 | 10 | 16 | 36
    III | 15 | 12 | 9 | 36
    IV | 0 | 0 | 0 | 0
    Subject does not have heart failure | 6 | 7 | 8 | 21
    Missing | 0 | 0 | 1 | 1
Minnesota Living with Heart Failure Questionnaire (MLWHF) [Mean (Standard Deviation); unit: units on a scale] — Minnesota Living with Heart Failure Questionnaire (MLWHF) is a health-related quality of life questionnaire. The scale ranges from 0 to 105. In particular, the lower the score the better is the patient's quality of life.
  units on a scale | 21 (25) | 29 (26) | 32 (29) | 28 (27)

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End Diastolic Volume (LVEDV)
Description: Left ventricular end diastolic volume (LVEDV) was measured by echocardiogram. Change was measured as Month 18 LVEDV minus baseline LVEDV.
  Per protocol, change in LVEDV is compared between Pooled Pacing (Single site + Dual Site) and Control.
Time Frame: Baseline - 18 Month Follow Up Visit
Population: The primary analysis cohort for the main objective of this study (Change in Left Ventricular End Diastolic Volume) required a subject to be randomized, and if randomized to Dual Site or Single Site, the subject must have had a successful implant. Moreover, only subjects with observed LVEDV at baseline and 18-month follow-up visit are included.
Measure: Mean (95% Confidence Interval); unit: mL
Groups:
- Pooled Pacing: Subjects successfully implanted with a CRT-D device (either single or dual pacing).
- Control: Subjects randomized to the group that did not have a device implanted and was managed according to conventional medical management.
Arm/Group | Pooled Pacing | Control
Number analyzed (Participants) | 64 | 34
mL | 16.4 [8.9 to 23.9] | 15.8 [5.5 to 26.2]

2. Secondary Outcome: Safety of Implanting a Cardiac Resynchronization Therapy With Defibrillator (CRT-D) Device Within 10 Days of Myocardial Infarction (MI), as Measured by the Rate of Reported Adverse Events
Description: Survival estimates at 18 months post-implant for time to first following events: (a) System Related Adverse Event (b) System Related Complication (c) Procedure Related Adverse Event (d) Procedure Related Complication and (e) System Related or Procedure Related Complication.
Time Frame: 18 months post-implant
Population: Only subjects with attempt implant are included. Therefore, subjects from the Control Arm are not included.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Single Site Pacing | Dual Site Pacing
Number analyzed (Participants) | 38 | 38
survival probability
  System-Related Adverse Event | 0.59 [0.41 to 0.73] | 0.68 [0.50 to 0.80]
  System Related Complication | 0.86 [0.70 to 0.94] | 0.87 [0.71 to 0.94]
  Procedure Related Adverse Event | 0.57 [0.40 to 0.71] | 0.66 [0.48 to 0.78]
  Procedure Related Complication | 0.84 [0.68 to 0.92] | 0.84 [0.68 to 0.93]
  System Related or Procedure Related Complication | 0.79 [0.62 to 0.89] | 0.82 [0.65 to 0.91]

3. Secondary Outcome: Frequency of Hospitalization for Cardiovascular Events
Description: Number of hospitalizations related to cardiovascular events.
Time Frame: Baseline - 18 Month Follow Up Visit
Population: Subject was randomized, and if randomized to Dual Site or Single Site, the subject must have had a successful implant.
Measure: Number; unit: participants
Groups:
- Single Site Pacing: Subjects randomized to the group that were successfully implanted with a CRT-D that delivers pacing via the Left Ventricular lead.
- Dual Site Pacing: Subjects randomized to the group that were successfully be implanted with a CRT-D that delivers pacing via the Left Ventricular and Right Ventricular lead.
Arm/Group | Single Site Pacing | Dual Site Pacing | Control
Number analyzed (Participants) | 38 | 37 | 45
participants
  0 | 27 | 22 | 30
  1 | 6 | 9 | 11
  2 | 3 | 3 | 0
  3 | 1 | 1 | 3
  4 | 0 | 0 | 0
  5 | 1 | 1 | 0
  6 | 0 | 0 | 0
  7 | 0 | 0 | 0
  8 | 0 | 1 | 0
  9 | 0 | 0 | 1

4. Secondary Outcome: Change in New York Heart Association (NYHA) Functional Class
Description: The New York Heart Association (NYHA) score classifies patients' heart failure according to the severity of their symptoms. In particular, Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Unable to carry on any physical activity without discomfort.
  NYHA change from baseline to 18-month visit. If a subject improved by one NYHA class or more (e.g. NYHA IV to NYHA II, or NYHA III to NYHA I, etc) from the baseline visit, the subject was classified as "Improved". Similarly for "Worsened" (e.g. subject does not have heart failure to NYHA I, NYHA I to NYHA II, etc.). If the subjects' NYHA Class is not different than baseline, then the subject was classified as "No Change".
  Per protocol, change in NYHA is compared between Pooled Pacing (Single site + Dual Site) and Control.
Time Frame: Baseline - 18 Month Follow Up Visit
Population: Subject was randomized, and if randomized to Dual Site or Single Site, the subject must have had a successful implant. Moreover, only subjects with observed NYHA at baseline and 18-month follow-up visit are included.
Measure: Number; unit: participants
Arm/Group | Pooled Pacing | Control
Number analyzed (Participants) | 68 | 33
participants
  Improved | 26 | 13
  No Change | 25 | 10
  Worsened | 17 | 10

5. Secondary Outcome: Change in 6-minute Walk Test Distance
Description: Change in 6-minute hallwalk distance from 1-month visit to the 18-month visit.
  Change is defined as month 18 minus baseline.
  Per protocol, change in 6-minute walk test distance is compared between Pooled Pacing (Single site + Dual Site) and Control.
Time Frame: 1 Month - 18 Month Follow Up Visit
Population: Randomized subjects, and if randomized to Dual Site or Single Site, the subject must have had a successful implant. Moreover, only subjects with observed 6-minute hallwalk distance at baseline and 18-month follow-up visits are included.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Pooled Pacing | Control
Number analyzed (Participants) | 63 | 28
meters | 37.6 [5.8 to 69.3] | 15.6 [-32.1 to 63.2]

6. Secondary Outcome: Change in Quality of Life
Description: Change in the Minnesota Living with Heart Failure (MNLWHF) questionnaire from baseline to the 18-month follow-up visit.
  Change is defined as month 18 minus baseline.
  Per protocol change in MNLWHF is compared between Pooled Pacing (Dual Site + Single Site) and Control.
Time Frame: Baseline - 18 Month Follow Up Visit
Population: Randomized subjects, and if randomized to Dual Site or Single Site, the subject must have had a successful implant. Moreover, only subjects with observed MNLWHF questionnaire score at baseline and 18-month follow-up visits are included.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pooled Pacing | Control
Number analyzed (Participants) | 69 | 32
units on a scale | 0.4 [-5.3 to 6.1] | -0.1 [-8.5 to 8.3]

7. Secondary Outcome: Incidence of Sudden Cardiac Death and Total Mortality
Description: Mortality rates (%) for the events (a) all-cause death and (b) sudden-cardiac death at 18 months post randomization. Calculated using Kaplan-Meier methods.
  Per protocol the comparison of mortality rates is between Pooled Pacing (Dual Site + Single Site) and Control.
Time Frame: 18 Months post-randomization
Population: Randomized subjects, and if randomized to Dual Site or Single Site, the subject must have had a successful implant.
Measure: Number (95% Confidence Interval); unit: percentage of subjects at risk
Arm/Group | Pooled Pacing | Control
Number analyzed (Participants) | 75 | 45
percentage of subjects at risk
  All-cause Death | 4.0 [1.3 to 12.0] | 4.7 [1.2 to 17.5]
  Sudden-cardiac Death | 1.4 [0.2 to 9.2] | 2.4 [0.3 to 16.1]

8. Secondary Outcome: Linear Association Between Change in LVEDV and Selected Clinical Characteristics; Including Peak Creatinine Phosphokinase (CPK), Peak Troponin, Lead Location, Time From MI Onset to Implant, and Change in LV Volumes.
Description: Linear association between change in LVEDV from baseline to 18-month visit (i.e. ΔLVEDV) and the following clinical characteristics were assessed: age, days from MI to implant, gender, hypertension, hyperlipidemia, diabetes, peak CPK, infarct location, LV electrode in acceptable place, and baseline LVEF. In order to assess these linear associations, linear regression models were fitted for each of these clinical characteristics (separately). In particular, each linear regression model had baseline LVEDV and the clinical characteristic as covariates, and ΔLVEDV was the response variable.
  Variables resulting in statistical significant (p<0.05) are reported.
Time Frame: Baseline - 18 Month Follow Up Visit
Population: All subjects randomized, and if randomized to Dual Site or Single Site, the subject must have had a successful implant. Moreover, only subjects with observed LVEDV at baseline and 18-month follow-up visit are included.
Measure: Mean (Standard Error); unit: regression coefficient
Groups:
- All Subjects: All subjects randomized in the study (either control, single pacing or dual pacing). For the patients randomized to single or dual site, only patients with successful implant are included.
Arm/Group | All Subjects
Number analyzed (Participants) | 98
regression coefficient
  Age | -0.75 (0.26)
  Days from MI to Implant* | -3.78 (1.64)
  Baseline LVEF | -0.87 (0.35)

ADVERSE EVENTS:
Arm/Group | Single Site Pacing | Dual Site Pacing | Control
Serious Adverse Events (participants affected / at risk) | 22/40 | 24/41 | 20/45
Other Adverse Events (participants affected / at risk) | 20/40 | 25/41 | 27/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Site Pacing (N=40) | Dual Site Pacing (N=41) | Control (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (5)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (2) | 3 (5)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (7) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 4 (6)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Decompensated Heart Failure (Cardiac disorders) | 2 (4) | 5 (13) | 6 (6)
Dresslers syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 2 (2)
Device infusion issue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device stimulation issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Implant site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lead dislodgement (General disorders) | 2 (3) | 4 (4) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 4 (4)
Undersensing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral myocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Site Pacing (N=40) | Dual Site Pacing (N=41) | Control (N=45)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Decompensated Heart Failure (Cardiac disorders) | 1 (1) | 3 (3) | 4 (5)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypogonadism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 3 (3) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3) | 2 (2)
Device alarm issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device capturing issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device electrical impedance issue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device infusion issue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (3) | 0 (0)
Device pacing issue (General disorders) | 4 (4) | 1 (1) | 0 (0)
Device stimulation issue (General disorders) | 8 (13) | 4 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Implant site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site scar (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lead dislodgement (General disorders) | 2 (2) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oversensing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 0 (0)
Phantom shocks (General disorders) | 0 (0) | 2 (2) | 0 (0)
Undersensing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Echinococciasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cardiac vein dissection (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Cardiac vein perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Biopsy skin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Echocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less